CLINICAL TRIAL: NCT03644758
Title: Assessment of the Quality of Sleep and Sleep Disorders Among the Professional and Volunteer Firefighters of Loire
Acronym: FIRESLEEP
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 18CH087; ANSM (Other: 2018-A01462-53)
Record Dates: First submitted 2018-08-22; First posted 2018-08-23 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Firefighter
Keywords: Firefighter; Sleep; Sleep disorders; Pittsburgh Sleep Quality Index (PSQI); Epworth Sleepiness Scale; Insomnia Severity Index (ISI); stop-BANG questionnaire
MeSH Terms: conditions — Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- professional and voluntary firefighter: Professional and voluntary firefighter in Service Departmental Fire and Rescue of Loire will be included. They will have to answer at the self-administrated questionnaires. It is composed of 5 parts: socio-demographic data and personal medical history, Pittsburgh Sleep Quality Index (PSQI), Epworth Sleepiness Scale, Insomnia Severity Index (ISI) and stop-BANG questionnaire.
  Interventions: Diagnostic Test: socio-demographic data and personal medical history; Diagnostic Test: Pittsburgh Sleep Quality Index (PSQI); Diagnostic Test: Epworth Sleepiness Scale; Diagnostic Test: Insomnia Severity Index (ISI); Diagnostic Test: stop-BANG questionnaire

INTERVENTIONS:
Diagnostic Test: socio-demographic data and personal medical history — Socio-demographic data and personal medical history is a self-administered questionnaire.
Diagnostic Test: Pittsburgh Sleep Quality Index (PSQI) — Pittsburgh Sleep Quality Index (PSQI) is a self-administered questionnaire. This score evaluates sleep disturbances.
Diagnostic Test: Epworth Sleepiness Scale — Epworth Sleepiness Scale is a self-administered questionnaire. This score evaluates excessive drowsiness.
Diagnostic Test: Insomnia Severity Index (ISI) — Insomnia Severity Index (ISI) is a self-administered questionnaire. This score evaluates insomnia severity.
Diagnostic Test: stop-BANG questionnaire — Stop-BANG is a self-administered questionnaire. This score evaluates Obstructive Sleep Apnea (OSA).

SUMMARY:
Studies have shown that schedules that most disrupt the normal circadian rhythm have the most harmful consequences. Firefighters positive for a sleep disorder have a higher risk of depression and anxiety; they report more traffic accidents, falling asleep during driving, and worth health felt. Furthermore, some studies suggest that sleep disorders are risk factors for cardiovascular disease. This activity is responsible of a worth quality of sleep that could induce a lower effectiveness of emergency response. The consequences of this schedules on sleep and health of French firemen have never been studied.

DETAILED DESCRIPTION:
In this context, the objective of this observational epidemiological study is to evaluate the quality of sleep of the firefighters of Loire.

ELIGIBILITY:
Inclusion Criteria:

* Any professional or voluntary firefighter active in Service Departmental Fire and Rescue of Loire or in retirement, and also the medical and paramedical staff of Service Departmental Fire and Rescue of Loire.
* Any fireman affiliated to a social security regime.
* Any fireman who has received information from the study and has agreed to participate in the study.

Exclusion Criteria:

* Any fireman unable to understand the study.
* Any fireman having a legal protection measure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Professional or voluntary firefighter will be included.
Sampling Method: Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2019-05-14 (Actual); Study Completion 2019-05-14 (Actual)

PRIMARY OUTCOMES:
sleep disturbances | September 2019
  Analyzed the percentage of firefighters with a score greater than 5 on the self-administrated questionnaire Pittsburgh Sleep Quality Index (PSQI) (Buysse and al., 1989).
  This score evaluates sleep disturbances.

SECONDARY OUTCOMES:
excessive drowsiness | September 2019
  Analyzed the percentage of firefighters totalizing a score of 10 or more during the self-realization of the Epworth Sleepiness Scale (Johns 1991).
  This score evaluates excessive drowsiness.
insomnia severity | September 2019
  Analyzed the percentage of firefighters totalizing a score of 10 on the auto-administrated questionnaire of Insomnia Severity Index (Bastien 2001).
  This score evaluates insomnia severity.
Obstructive Sleep Apnea (OSA) | September 2019
  Analyzed the percentage of firefighters with a high-risk of obstructive sleep apnea syndrome on the STOP-Bang questionnaire (Chung et al., 2012).
  This score evaluates the risk of doing an Obstructive Sleep Apnea (OSA).
status firefighter | September 2019
  Correlation between status firefighter (professional or voluntary firefighter) and the scores of Epworth Sleepiness Scale, Pittsburgh Sleep Quality Index (PSQI), Insomnia Severity Index (ISI) and stop-BANG.
number of years of professional practice | September 2019
  Correlation between number of years of professional practice as a firefighter and the scores of Epworth Sleepiness Scale, Pittsburgh Sleep Quality Index (PSQI), Insomnia Severity Index (ISI) and stop-BANG.
fire station | September 2019
  Correlation between fire station and the scores of Epworth Sleepiness Scale, Pittsburgh Sleep Quality Index (PSQI), Insomnia Severity Index (ISI) and stop-BANG.
exercise of another professional activity | September 2019
  Correlation between exercise of another professional activity and the scores of Epworth Sleepiness Scale, Pittsburgh Sleep Quality Index (PSQI), Insomnia Severity Index (ISI) and stop-BANG.
shift schedules 12 or 24 hours | September 2019
  Correlation between shift schedules 12 or 24 hours and the scores of Epworth Sleepiness Scale, Pittsburgh Sleep Quality Index (PSQI), Insomnia Severity Index (ISI) and stop-BANG.
family status | September 2019
  Correlation between shift family status and the scores of Epworth Sleepiness Scale, Pittsburgh Sleep Quality Index (PSQI), Insomnia Severity Index (ISI) and stop-BANG.
personal medical history | September 2019
  Correlation between personal medical history and the scores of Epworth Sleepiness Scale, Pittsburgh Sleep Quality Index (PSQI), Insomnia Severity Index (ISI) and stop-BANG.
number of interventions by guard | September 2019
  Correlation between number of interventions by guard and the scores of Epworth Sleepiness Scale, Pittsburgh Sleep Quality Index (PSQI), Insomnia Severity Index (ISI) and stop-BANG.
number of interventions by constraint | September 2019
  Correlation between number of interventions by constraint and the scores of Epworth Sleepiness Scale, Pittsburgh Sleep Quality Index (PSQI), Insomnia Severity Index (ISI) and stop-BANG.

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric ROCHE, PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No